CLINICAL TRIAL: NCT03765619
Title: Effects of Postoperative Aspirin on Ankle Fracture Healing
Brief Title: Postoperative Aspirin and Ankle Fracture Healing
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ashish Shah, M.D., Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB-300002057
Record Dates: First submitted 2018-11-08; First posted 2018-12-05 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures | interventions — Aspirin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin (Experimental): 250 patients will be randomized to receive Aspirin postoperatively.
  Interventions: Drug: Aspirin
- Non-Aspirin (No Intervention): 250 patients will be randomized to not receive Aspirin postoperatively.

INTERVENTIONS:
Drug: Aspirin — 250 patients will be randomized to receive postoperative Aspirin.
  Arms: Aspirin

SUMMARY:
This study aims to identify if postoperative aspirin use leads to a delay in fracture healing. NSAIDs have long been avoided in the management of fractures, due to the belief that they may impair fracture healing. As aspirin is frequently prescribed for long-term management of various medical conditions, it is worth understanding if continuing to take aspirin during the process of fracture healing has a clinically significant effect on the rate of fracture healing.

DETAILED DESCRIPTION:
Despite any new clinical research on aspirin's effects on fracture healing, it is now being used more commonly in the setting of fracture due to its effectiveness as a means of VTE prophylaxis following major orthopedic surgery.5 Additionally, aspirin offers the benefit of acting as an analgesic and many patients are prescribed aspirin in the long-term management of various health conditions. With all of the potential therapeutic benefits of aspirin, it is worth understanding whether prescribing this medication following operative fracture repair may impose a risk of delayed fracture healing.

Patients undergoing surgical repair of ankle fractures at UAB who are deemed healthy enough for orthopedic surgery will be enrolled. Patients with multiple traumatic injuries, patients taking any type of blood-thinner medication, and patients taking aspirin prior to the start of the study will be excluded. No other exclusions will be made based on prior health conditions. There will be a group of patients that receives no aspirin and a group that does receive aspirin. Approximately 250 patients will be randomly assigned to each group.

Patients will be identified for potential enrollment based on their plan to undergo surgical repair of ankle fracture at UAB hospital during the IRB approval period. This study will follow patients following routine protocol for ankle fracture repair and follow-up. Patients will be randomized into a group that is prescribed aspirin (325 mg) post-operatively vs. not prescribed aspirin. Patients will be followed throughout their recovery process. Patients will be scheduled for follow-up appointments with the operating physician at 2 weeks, 6 weeks, 3 months, 6 months, and 1 year following surgery. Patients will be asked to give a pain score (scale 1-10) and complete an SF-12 functional outcomes survey at each follow-up appointment. In line with normal protocol following fracture repair, radiographs will also be taken at each follow-up appointment to monitor the progression of fracture healing.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* healthy enough for orthopedic surgery
* slated to undergo surgical repair of ankle fracture at UAB
* able to give consent All ankle fractures (lateral malleolus, medial malleolus, bimalleolar, trimalleolar, and proximal fibula) will be included in this study.

Exclusion Criteria:

* Under 18 years of age
* inability to give consent
* Pilon fractures
* Multiple traumatic fractures
* Known history of aspirin allergy
* History of severe reaction to aspirin
* History of bleeding disorder
* Other clear contraindication to being prescribed aspirin
* Taking blood-thinning medications (heparin, apixaban, etc)
* Taking aspirin prior to the start of the study

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Ankle Fracture Healing | 0 - 12 months following surgery
  Union Rates of Ankle Fractures postoperatively as assessed clinically and radiographically. X-rays will be taken at each postoperative visit.

SECONDARY OUTCOMES:
Functional Outcomes | 0 - 12 months following surgery
  Patients will complete an Short Form-12 functional outcomes survey at each follow-up appointment, which is a health outcomes scale that includes assessment of general health, physical function, pain, social function, and mental health. Scores are combined to give Physical Health Composite Scores and Mental Health Composite Scores. Scale is 0 - 100, with lower scores indicating worse outcomes, and higher scores indicating better outcomes.
Visual Analog Scale for Pain | 0 - 12 months following surgery
  Patients will disclose their pain level using the Visual Analog Scale, which measures pain on a scale of 0 - 100, with 0 indicating no pain and 100 indicating severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Highland Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No